CLINICAL TRIAL: NCT00507585
Title: A Phase I Study of Hepatic Arterial Infusion of Oxaliplatin in Combination With Systemic Fluorouracil, Leucovorin and Avastin for Patients With Advanced Solid Tumors Metastatic to the Liver
Brief Title: Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, Leucovorin, and Avastin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0160
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Liver Cancer; Advanced Solid Tumors
Keywords: Liver Cancer; Liver metastases; Metastatic advanced solid tumors; Advanced solid tumors metastatic to the liver; Hepatic Arterial Infusion; Intra-arterial hepatic oxaliplatin; Fluorouracil; 5-FU; Adrucil; Efudex; 5-fluorouracil; Avastin; Leucovorin; Oxaliplatin; Bevacizumab
MeSH Terms: conditions — Liver Neoplasms | interventions — Fluorouracil; Bevacizumab; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxaliplatin + Fluorouracil + Leucovorin + Avastin (Experimental)
  Interventions: Drug: Fluorouracil; Drug: Avastin; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Fluorouracil — 300 mg/m^2 IV over 10 Minutes, then 600 mg/m^2 IV over 22 Hours repeated every 3 weeks (1 Cycle).
  Other Names: 5-FU; Adrucil; Efudex; 5-fluorouracil
Drug: Avastin — 10 mg/m^2 IV Over 90 Minutes repeated every 3 weeks (1 Cycle).
  Other Names: Bevacizumab
Drug: Leucovorin — 200 mg/m^2 IV Over 2 Hours repeated every 3 weeks (1 Cycle).
Drug: Oxaliplatin — 60 mg/m^2 IV Over 2 Hours repeated every 3 weeks (1 Cycle).

SUMMARY:
PRIMARY:

* To determine the toxicity and tolerability of intra-arterial hepatic oxaliplatin every three weeks administered in combination with systemic intravenous Fluorouracil, Leucovorin and bevacizumab to patients with advanced solid tumors metastatic to the liver.

SECONDARY:

* To document in a descriptive fashion the antitumor efficacy of this combination regimen.
* To evaluate the feasibility and accuracy of an alternate radiographic assessment tool and compare with available tumor markers and RECIST guidelines.
* To estimate in a descriptive fashion the development of extrahepatic tumor recurrences.

DETAILED DESCRIPTION:
Oxaliplatin is designed to interfere with the growth of cancer cells (which slows their growth and spreading), eventually destroying them.

5-fluorouracil is designed to interfere with the growth of cells that reproduce rapidly.

Leucovorin is designed to strengthen the effect of 5-fluorouracil by reducing tumor cell resistance to the 5-fluorouracil.

Bevacizumab is designed to interfere with blood flow to your tumors, which may cause tumors to be "starved" of the oxygen and nutrients they need to grow.

Before you can start on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have your complete medical history recorded and a physical exam, including measurement of your vital signs (blood pressure, temperature, breathing rate, and heart rate). You will have a neurological evaluation (a test to evaluate your strength and nerve functioning). You will have blood drawn (about 1 teaspoon or less) and urine collected for routine tests. Women who are able to have children must have a negative urine pregnancy test.

If you are found to be eligible to take part in this study, you will be hospitalized to receive the study drug combination. On the day of your admission to the hospital, you will have a catheter in your hepatic artery placed in your right groin. After your catheter has been placed, you will receive the study drugs. The catheter will be placed and removed during each cycle. A catheter is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your physician will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure.

You must lay in bed for the entire time that the catheter is in place. In some cases, the catheter will be removed immediately after your chemotherapy is complete. In some cases, the catheter may remain in overnight. Therefore, you must remain in bed until the catheter is removed.

During each cycle (on Days 1 and 2), you will receive 5-fluorouracil by vein continuously over 24 hours, leucovorin by vein over 1 hour, oxaliplatin by your hepatic artery over 2 hours, and bevacizumab by vein (only on Day 1) over about 1 1/2 hours. This study drug combination will be repeated about every 3 weeks, which is considered 1 cycle (about every 21 days).

To learn the highest tolerable dose of oxaliplatin when given in combination with the other study drugs, there will be a dose escalation process that will go as follows. The dose of oxaliplatin that you receive will depend on when you are enrolled in this study. The dose of the other 3 study drugs that you receive will be the same for each participant on this study. At first, 6 participants will be enrolled at the first dose level of oxaliplatin. If their disease does not get worse and no intolerable side effects occur, there will be another 6 patients enrolled at the next higher dose level. This dose escalation process will continue in this way until 8 dose levels have been reached without intolerable side effects occurring.

You will have blood drawn (about 2 teaspoons each) for blood counts and liver function tests before each dose of the study drug combination. This is so your doctor can check the safety of the drug combination. You will also have blood drawn (about 2 teaspoons each) before each cycle. The doctor will evaluate your disease and health before you receive the study drugs. Your tumors will be evaluated by the imaging scans (such as computed tomography [CT] and magnetic resonance imaging [MRI]) needed for your type of cancer. Imaging scans will be performed every 2 cycles.

You may continue to receive the study drug combination indefinitely as mentioned above unless your disease gets worse or you experience any intolerable side effects. If your disease gets worse or you experience any intolerable side effects, you will be removed from this study.

If your participation ends for any reason on this study (such as those mentioned above), you will have imaging scans (CT and MRI) to see if your tumors are growing or shrinking. You will have blood drawn (about 3 teaspoons) for routine tests. These end-of-study tests can be performed at your regular doctor's office, and the results will be sent to the study's research staff.

This is an investigational study. Oxaliplatin is authorized by the FDA for systemic use only. (Systemic therapies affect the body as a whole.) Giving oxaliplatin directly into the liver is investigational. 5-fluorouracil, leucovorin, and bevacizumab are FDA-approved for treatment of colorectal cancer. The use of these drugs in combination is authorized by the FDA for use in research only. Bevacizumab is not FDA-approved for all cancer types included in this study. Up to 163 patients will take part in this study. All patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed metastatic advanced solid tumors involving the liver.
2. Pediatric patients eligible at the discretion of the primary investigator.
3. Performance status ECOG 0-2 (Capable of all self care but unable to to carry out any work activities).
4. Adequate renal function (Serum Creatinine </= 2.0 mg/dL) or a calculated creatinine clearance greater than 60 mL/min.
5. Hepatic function as follows: In treatment arm 1: Total Bilirubin </= 3 mg/dL, AST </= 5 times upper normal reference value, or ALT </= 5 times upper normal reference value). In treatment arm 2: Total bilirubin >3 mg/dL. If bilirubin >/= 5 mg/dL, fluorouracil (5FU) dose will be omitted.
6. Adequate bone marrow function (ANC >/=1500 cells/uL; PLT >/= 100,000 cells/uL).
7. At least three weeks from previous immunotherapy, chemotherapy or radiotherapy before day of HAI infusion and recovery from any associated toxicities to less or equal to Grade 1.
8. All females in childbearing age MUST have a negative serum HCG test unless prior hysterectomy or menopause (defined as age above 55 and six months without menstrual activity). Patients should not become pregnant or breast feed while on this study. Sexually active patients should use effective birth control.
9. Ability to fully read, comprehend, and sign informed consent forms.

Exclusion Criteria:

1. Clinical or radiographic evidence of ascites.
2. Pregnant females.
3. Inability to complete informed consent process and adhere to protocol treatment plan and follow-up requirements.
4. Grade 2 Peripheral Neuropathy (CTC V3.0: Sensory alteration interfering with function but not interfering with ADL)
5. Serious or non-healing wound, ulcer or bone fracture.
6. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days.
7. Invasive procedures defined as follows; Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1 therapy, Anticipation of need for major surgical procedures during the course of the study, Core biopsy within 7 days prior to D1 of therapy.
8. Patients receiving any other investigational agents.
9. Patients with bleeding diathesis (clinical bleeding, prothrombin time =/> 1.5 X upper institutional normal value, INR =/> 1.5, activated partial thromboplastin time aPTT =/> 1.5 X upper institutional normal value), active gastric or duodenal ulcer.
10. Uncontrolled systemic vascular hypertension (Systolic blood pressure > 140 mmHg, Diastolic Blood Pressure > 90 mmHg).
11. Urine protein should be screened by dipstick or urine analysis. For proteinuria > 1+ or urine protein:creatinine ratio > 1.0, a 24-hour urine protein should be obtained and the level should be < 1000 mg for patient enrollment.
12. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
13. Patients with clinically significant cardiovascular disease: History of CVA within 6 months, myocardial infarction or unstable angina within 6 months, New York Heart Association Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, unstable angina pectoris, clinically significant peripheral vascular disease
14. Patients with history of bleeding CNS metastasis will be excluded from the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To study the highest tolerable dose of oxaliplatin used in combination with 5-fluorouracil, leucovorin, and Avastin® (bevacizumab) for patients with advanced cancer that has spread to the liver. | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia M. Tsimberidou, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org